CLINICAL TRIAL: NCT05824468
Title: A Phase II Trial of Zimberelimab Plus Lenvatinib After Progression on Prior Immune Checkpoint Inhibitors in Patients With Advanced Cervical Cancer
Brief Title: Zimberelimab Plus Lenvatinib After Progression on Prior Immune Checkpoint Inhibitors for Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-098-01
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Cervical Cancer; Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — zimberelimab; spartalizumab; lenvatinib; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Intervention Model Description: Drug: Zimberelimab, Drug: Lenvatinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zimberelimab + Lenvatinib (Experimental): Safety run-in phase A dose de-escalation schedule is used in this phase. Dose Level 1: zimberelimab 240 mg administered intravenously on day 1 and lenvatinib 16 mg administered orally once daily on a 21-day treatment cycle. If ≥2/6 patients experience a DLT, we will de-escalate to Dose Level 2: zimberelimab 240 mg administered intravenously on day 1 and lenvatinib 12 mg administered orally once daily on a 21-day treatment cycle. Approximately 3-12 patients will be enrolled in the safety run-in phase.
  Expansion phase The expansion stage will begin once the RP2D of lenvatinib have been determined in the safety run-in phase in order to assess antitumor activity of zimberelimab and lenvatinib combination. In expansion stage, zimberelimab 240 mg administered intravenously and lenvatinib PR2D will be administered.
  Interventions: Drug: Zimberelimab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Zimberelimab — Injectable solution
  Other Names: Anti-PD-1 antibody
Drug: Lenvatinib — Capsule
  Other Names: Tyrosine Kinase Inhibitor

SUMMARY:
Although immune checkpoint inhibitors (ICIs) provide a durable response in multiple tumor types, relapse occurs in most patients with solid tumor. However, the benefits of retreatment with ICIs remains controversial. In some studies, retreatment with ICIs has exhibited encouraging efficacy in patients with solid tumors, particularly in melanoma, and non-small cell lung cancer (NSCLC). In this single arm phase 2 trial, we aimed to evaluate the efficacy and safety of the combination of anti-PD1 antibody (zimberelimab) and lenvatinib in patients with advanced cervical cancer who progressed on or after prior ICIs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF).
2. Has histologically confirmed diagnosis of metastatic, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy.
3. Has progressed on at least one line of platinum-based systemic therapy. Note: Prior adjuvant therapy is NOT counted as a systemic chemotherapeutic regimen for management of recurrent, persistent or metastatic cervical cancer; adjuvant therapy includes cisplatin given concurrent with primary radiation therapy and adjuvant chemotherapy given following the completion of concurrent chemotherapy and radiation therapy. However, adjuvant chemotherapy could be counted as one prior regimen in patients who had recurrence during or within 6 months of completion of therapy.
4. Has progressed on or after treatment of prior immune checkpoint inhibitors (ICIs), with the exposure of ICIs more than 6 months.
5. Age ≥ 18 years and ≤ 75 years.
6. Has measurable disease per RECIST v1.1; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded as ≥ 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI); a lymph node must be ≥ 15 mm in short axis. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Life expectancy exceeds 3 months.
9. Has adequate organ function as defined by the following criteria:

   * Absolute neutrophil count (ANC) (≥1.5×109/L), hemoglobin of ≥90 g/L, platelets ≥100 ×109/L
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN (however, patients with known liver metastasis who have AST or ALT level ≤ 5 × ULN may be enrolled)
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula)
10. Females of childbearing potential should have a negative serum or urine pregnancy test prior to receiving the first dose of study treatment; and should be willing to use one acceptable contraception (i.e., oral contraceptives, condoms, intrauterine devices [IUDs]) throughout the period of taking study treatment and for at least 6 months after the last dose of study drug(s).

Exclusion Criteria:

1. Histologic types of carcinoma other than squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma.
2. Known or suspected allergy to any of study drugs.
3. Prior exposure to small molecule anti-angiogenic agent.
4. Has an active autoimmune disease requiring systemic therapy (i.e., with use of disease modifying drugs, corticosteroids or immunosuppressive drugs) in past 2 years. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permitted.
5. Concurrent medical condition requiring the use of systemic steroid therapy (dose > 10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy within 2 weeks prior to the first dose of study intervention.
6. Has an active infection requiring systemic therapy.
7. Any unresolved toxicities from prior therapy, greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with exception of alopecia and anemia.
8. Recieved major surgery with 28 days before the first medication or has serious nonhealing wound, or ulcer.
9. Clinically significant cardiovascular diseases, including but not limited to congestive heart failure (New York heart association [NYHA] class > 2), unstable or severe angina, severe acute myocardial infarction within 6 months before enrollment, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.
10. Hypertension that can not be well controlled through antihypertensive drugs (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mmHg).
11. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
12. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
13. Coagulation abnormalities (INR > 2.0, PT > 16s), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
14. Has known active central nervous system metastases.
15. History of another malignancy in the previous 3 years, with a disease-free interval of <3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy. Patients who have undergone a bone marrow or stem-cell transplant for any malignancy are excluded.
16. Has a known history of immunodeficiency including human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease.
17. Has known active hepatitis B disease (hepatitis B virus [HBV] DNA ≥ 1×104/ml) or hepatitis C disease (hepatitis C virus [HCV] RNA ≥ 1×103/ml).
18. Has received a live vaccine within 30 days prior to the first dose of trial treatment. Note: Injection of inactivated viral vaccines against seasonal influenza are allowed.
19. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | the first 21 days of treatment
  MTD is defined as the highest dose level at which no more than 1 out of 6 subjects experiences a dose limiting toxicities (DLT) during the first cycles.
Recommended Phase 2 dose (RP2D) | the first 21 days of treatment
  Determine the RP2D of lenvatinib
Response Rate (ORR) | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | from the first drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD.
Duration of response (DOR) | from the first drug administration up to two years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first.
Overall survival (OS) | from the first drug administration up to 2 years
  Time from the date of first study treatment administration to the date of death due to any cause.
Safety and tolerability | up to 90 days after last study treatment administration
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

OTHER OUTCOMES:
Biomarkers associated with the response to zimberelimab plus lenvatinib | Samples taken prior to the first dose of drug, Cycle 3 and at progression
  Exploration of biomarkers that predict the efficacy of retreatment of anti-PD-1 antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Cetntre, Guangzhou, China